CLINICAL TRIAL: NCT04337658
Title: A Phase 3, Randomized, Multicenter, Open-Label Study to Compare the Efficacy and Safety of Anti-HER2 Therapy Plus Fulvestrant or Capecitabine in First-line Treatment of Women With HR+, HER2+, Non-visceral Metastases, Stage IV Breast Cancer
Brief Title: Anti-HER2 Therapy + Fulvestrant/Capecitabine in Women With HR+, HER2+, Non-visceral Metastases Stage IV Breast Cancer
Acronym: FAVOR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, xuexin he, Principal Investigator, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAVOR
Record Dates: First submitted 2020-01-11; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: HER2-positive Breast Cancer
Keywords: breast cancer; hormone receptor positive; human epidermal growth factor receptor 2 positive; non-visceral metastases; fulvestrant; capecitabine; trastuzumab; pertuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Fulvestrant; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trastuzumab± Pertuzumab+ Fulvestrant (Experimental): Pertuzumab(Perjeta): Participants will receive 840 milligrams (mg) loading dose of pertuzumab, followed every 3 weeks thereafter by a dose of 420 mg via intravenous (IV) infusion until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. It depends on the patient's choice.
  Trastuzumab(Herceptin): Participants will receive trastuzumab (8 mg/kg loading dose for Cycle 1, followed by 6 mg/kg for subsequent cycles) administered by IV infusion every 3 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Fulvestrant(Faslodex): 500mg intramuscular injections at day 1, 15, 28 and every 4 weeks thereafter
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Fulvestrant
- Trastuzumab± Pertuzumab+ Capecitabine (Active Comparator): Pertuzumab(Perjeta): Participants will receive 840 milligrams (mg) loading dose of pertuzumab, followed every 3 weeks thereafter by a dose of 420 mg via intravenous (IV) infusion until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. It depends on the patient's choice.
  Trastuzumab(Herceptin): Participants will receive trastuzumab (8 mg/kg loading dose for Cycle 1, followed by 6 mg/kg for subsequent cycles) administered by IV infusion every 3 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Capecitabine: 1000mg/m2 orally Bid on day 1 to day 14 every 3 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Capecitabine

INTERVENTIONS:
Drug: Pertuzumab — Participants will receive 840 milligrams (mg) loading dose of pertuzumab, followed every 3 weeks thereafter by a dose of 420 mg via intravenous (IV) infusion until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Other Names: Perjeta
Drug: Trastuzumab — Participants will receive trastuzumab (8 mg/kg loading dose for Cycle 1, followed by 6 mg/kg for subsequent cycles) administered by IV infusion every 3 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Other Names: Herceptin
Drug: Fulvestrant — 500mg intramuscular injections at day 1, 15, 28 and 4 weeks thereafter
  Other Names: Faslodex
  Arms: Trastuzumab± Pertuzumab+ Fulvestrant
Drug: Capecitabine — 1000mg/m2 orally Bid on day 1 to day 14 every 3 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Other Names: Xeloda
  Arms: Trastuzumab± Pertuzumab+ Capecitabine

SUMMARY:
The purpose of this study is to evaluate the effectiveness of anti-HER2 therapy plus Fulvestrant or Capecitabine in women with hormone receptor positive (HR+), human epidermal growth factor receptor 2 positive (HER2+), non-visceral metastases, stage IV breast cancer.

DETAILED DESCRIPTION:
This is a prospective, randomized, 2-arm, multicenter study to compare the safety and efficiency of anti-HER2 therapy (Trastuzumab ± Pertuzumab) plus fulvestrant versus anti-HER2 therapy (Trastuzumab ± Pertuzumab) plus capecitabine in women with hormone receptor positive (HR+), human epidermal growth factor receptor 2 positive (HER2+), non-visceral metastases, stage IV breast cancer. Subjects will be randomized into one of two treatment arms. Arm A subjects will receive the anti-HER2 therapy plus fulvestrant. Arm B subjects will receive the anti-HER2 therapy plus capecitabine. The use of Pertuzumab depends on patients' choices.

ELIGIBILITY:
Inclusion Criteria:

1. Patients provided written informed consent
2. Postmenopausal or premenopausal or perimenopausal women aged 18-75 years:

   1. ≥60 years, or bilateral ovariectomy was previously performed, or
   2. <60 years, natural postmenopausal status (defined as a continuous period of at least 12 months following spontaneous cessation without other pathological or physiological causes), estrogen (E2) and follicle-stimulating hormone (FSH) are present at postmenopausal levels
   3. Premenopausal or perimenopausal women, willing to receive luteinizing hormone (LHRH) stimulation during the study
3. Histologically or cytologically confirmed HR-positive (ER/PR≥10%), HER2-positive (IHC 3+ or ISH+) breast cancer
4. At least one measurable non-visceral metastatic lesion (liver, lung, pleura, pericardium, peritoneum, kidney, adrenal, brain or leptomeningeal metastases are excluded), HR-positive (ER/PR≥10%), HER2-positive (IHC 3+ or ISH+), (≥10 mm on T1-weighted, gadolinium-enhanced MRI) (RECIST v1.1)
5. Previous treatment with HER2 inhibitors to be discontinued prior to first study treatment administration (at least 14 days for trastuzumab and other antibodies, at least 7 days for lapatinib)
6. Previous chemotherapy, biological or target therapy to recurrent or metastatic disease are not allowed; Previous radiotherapy allowed, but radiotherapy must have been discontinued at least 14 days prior to first study treatment administration.
7. Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2
8. Life expectancy > 24 weeks
9. left ventricular ejection fraction (LVEF) of 50% or higher at baseline (within 42 days before randomization)
10. Previous adjuvant chemotherapy treatment is allowed
11. Previous adjuvant trastuzumab treatment is allowed
12. Hormone therapy must have been discontinued at least 1 month prior to recruitment
13. Patients with good compliance
14. Patients must have recovered to baseline condition or to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade = 1 from any acute CTCAE v. 5.0 grade =2 side effects of previous treatments
15. Without infection of human immunodeficiency virus (HIV) on central laboratory assay results prior to randomization
16. Alanine aminotransferase (ALT) </= 2.5 × the upper limit of normal (ULN), Aspartate aminotransferase (AST) </= 2.5 × ULN prior to randomization
17. Total bilirubin (TBIL) </= 1.25 × ULN
18. Alkaline phosphatase (ALK) </= 2.5 × ULN
19. Gamma glutamyl transpeptidase (GGT) </= 2.5 × ULN
20. Serum total bilirubin (TBil) </= 1.5 × ULN
21. Serum creatinine (Scr) </= 1.5 × ULN
22. WBC >/= 3×109/L, Blood neutrophil count >/= 1×109/L, Platelet count >/= 100×109/L, HB >/= 9 g/dL
23. Albumin >/= 30g/L
24. Women of child-bearing age who had a negative serum pregnancy test (within 14 days before randomization) should take effective contraceptive measures

Exclusion Criteria:

1. Primary and metastatic lesion lack of histological or cytological confirmation of HR-positive (ER/PR≥10%), HER2-positive (IHC 3+ or ISH+)
2. Breast cancer with visceral metastases (liver, lung, pleura, pericardium, peritoneum, kidney, adrenal, brain or leptomeningeal metastases)
3. Inflammatory breast cancer
4. Having a life-threatening metastatic visceral disease, defined as extensive liver damage or brain or leptomeninges damage (past or present) or symptomatic pulmonary lymphatic diffusion. Patients with discrete pulmonary parenchyma metastasis were eligible if the investigators determined that their respiratory function was not significantly impaired by the disease.
5. Disease progression or recurrence within 12 months after neo/adjuvant endocrine therapy
6. Unable to tolerate endocrine therapy, including those who with symptoms, who have spread to the viscera, and who are at risk for short-term life-threatening complications (including uncontrolled thorax, pericardium, or abdominal cavity exudation, pulmonary lymphangitis, and more than 50% liver damage).
7. CT or MRI confirmed the presence of brain or leptomeningeal metastases.
8. Any other current malignancy or malignancy diagnosed within the past five years (other than breast cancer, carcinoma in situ of the cervix, skin basal cell carcinoma or squamous cell carcinoma), unless radical treatment is performed and there is no evidence of recurrence or metastasis within the last 5 years.
9. Non- visceral metastatic lesions cannot be evaluated by RECIST v1.1
10. Active infection with human immunodeficiency virus (HIV) prior to first study treatment administration.
11. History of participating any other clinical trials within 30 days prior to randomization
12. Known hypersensitivity (Grade 3 or 4) to Pertuzumab, Trastuzumab, Fulvestrant or Capecitabine or the excipients of any of the trial drugs
13. Pregnancy or lactation
14. Uncontrolled illnesses including symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia requiring therapy, myocardial infarction within the past 6 months, or active infection
15. severe pulmonary and renal disease
16. Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)
17. Legal incompetence or limitation.
18. Considered unable to complete the study or sign the informed consent due to a medical or mental disorder by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to approximately 2 years
  Progression-free survival (PFS) was defined as the time from randomization to first occurrence of progressive disease (PD), as determined by the investigator using RECIST v1.1, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to approximately 2 years
  Overall survival (OS) was defined as the time from randomization to death from any cause.
Clinical Benefit Rate (CBR) | up to approximately 2 years
  Clinical Benefit Rate (CBR) is estimated by dividing the number of patients with CR, PR, or SD (for patients with measurable disease) ≥ 24 weeks from randomization.
Duration of Clinical Benefit (DOCB) | up to approximately 2 years
  DOCB was defined as the time from randomization to first occurrence of progressive disease (PD), as determined by the investigator using RECIST v1.1, or death from any cause, whichever occurred first (only for patients of CB)
Safety:Type incidence and severity (as graded by NCI CTCAE v 5.0) | up to approximately 2 years
  Seriousness and attribution to the study medications of AEs

CONTACTS AND LOCATIONS:
Overall Officials: Xuexin He, MD, Principal Investigator — The Second Affiliated Hospital of Zhejiang University School of Medicine (SAHZU); Jiajia Huang, MD, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Second Affiliated Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang